CLINICAL TRIAL: NCT03958747
Title: A Pilot Study Using Ultrasound for the Detection of Oxaliplatin-Induced Peripheral Neuropathy
Brief Title: Ultrasound for the Detection of Oxaliplatin-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00059662; P30CA012197 (NIH); WFBCCC 97219 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms | interventions — Blood Specimen Collection; Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound (Experimental): Undergo peripheral nerve ultrasound
  Interventions: Diagnostic Test: Ultrasound - Serial and Tibial Nerve; Procedure: Skin Biopsy; Other: Abbreviated Neurologic Exam; Other: Blood draw; Diagnostic Test: Nerve Conduction Study; Other: QLQ-CIPN20 Questionnaire Administration

INTERVENTIONS:
Diagnostic Test: Ultrasound - Serial and Tibial Nerve — Participants will undergo a serial and tibial nerve ultrasound
Procedure: Skin Biopsy — Two skin biopsies will be obtained as 4.0 mm punch biopsies at distal end of leg in sural nerve territory (10 cm above lateral malleolus) and from the thigh
Other: Abbreviated Neurologic Exam — Exam to include strength assessment of the tibialis anterior and gastrocnemius and deep tendon reflex exam of the Achilles on the limb to be examined by nerve conduction velocity and ultrasound.
Other: Blood draw — 12 ml blood sample will be taken
Diagnostic Test: Nerve Conduction Study — Sural and tibial nerve assessments
Other: QLQ-CIPN20 Questionnaire Administration — Self-reported neuropathy scoring questionnaire completed same day as blood draw.

SUMMARY:
This pilot clinical trial studies how well ultrasound works in detecting oxaliplatin-induced neuropathy in patients with gastrointestinal cancer. Ultrasound may work better in diagnosing and detecting neuropathy in gastrointestinal cancer patients treated with the chemotherapy drug called a oxaliplatin.

DETAILED DESCRIPTION:
Primary Objectives

I. To compare tibial motor nerve ultrasound cross-sectional area between oxaliplatin-induced peripheral neuropathy patients and historical data among healthy adults.

Secondary Objective

I. To compare sural sensory nerve ultrasound cross-sectional area between oxaliplatin-induced peripheral neuropathy patients and historical data among healthy adults.

II. To determine if the above changes in nerve cross-sectional area correlate with nerve conduction study changes in the same oxaliplatin-induced peripheral neuropathy patients.

III. To determine if the above changes in nerve cross-sectional area correlate with changes on a self-reported neuropathy scale (QLQ-CIPN20) in the same oxaliplatin-induced peripheral neuropathy patients.

IV. To determine if the above changes in nerve cross-sectional area correlate with intraepidermal nerve fiber density changes on skin biopsy in the same oxaliplatin-induced peripheral neuropathy patients.

Exploratory Objectives I. To assess activated mast cells in skin biopsies in oxaliplatin-induced peripheral neuropathy patients in relation to severity of symptoms and above findings.

II. To assess serum inflammatory markers in oxaliplatin-induced peripheral neuropathy patients in relation to severity of symptoms and above findings.

III. Exploratory Cohort (Oxaliplatin-induced peripheral neuropathy, OIPN) Objectives

IV. To compare tibial motor nerve ultrasound cross-sectional area between oxaliplatin-induced peripheral neuropathy patients and historical data among healthy adults and OIPN patients

V. To compare sural sensory nerve ultrasound cross-sectional area between oxaliplatin-induced peripheral neuropathy patients and historical data among healthy adults and oxaliplatin-induced peripheral neuropathy patients

VI. To determine if the above changes in nerve cross-sectional area correlate with nerve conduction study changes in the same oxaliplatin-induced peripheral neuropathy patients

VII. To determine if the above changes in nerve cross-sectional area correlate with changes on a self-reported neuropathy scale (QLQ-CIPN20) in the same oxaliplatin-induced peripheral neuropathy patients

VIII. To determine if the above changes in nerve cross-sectional area correlate with intraepidermal nerve fiber density changes on skin biopsy in the same oxaliplatin-induced peripheral neuropathy patients

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal cancer
* Colorectal cancer (any stage)
* Previously or currently receiving oxaliplatin -based chemotherapy.
* Clinical symptoms of peripheral neuropathy noted in medical record and suspected to be secondary to oxaliplatin -based therapy.
* Ability and willingness to understand and sign an informed consent.

Exclusion Criteria:

* Self-reported or documented history of pre-existing peripheral neuropathy prior to initiation of oxaliplatin chemotherapy.
* Unable to provide history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Tibial Nerve Cross-Sectional Area Comparison | Up to 30 days
  Tibial nerve cross-sectional area determined by ultrasound in oxaliplatin-induced peripheral neuropathy patients will be transformed to compare to historical data previously collected from healthy adults and oxaliplatin-induced peripheral neuropathy patients using analysis of variance (ANOVA).

SECONDARY OUTCOMES:
Sural Nerve Cross-Sectional Area Comparison | Up to 30 days
  Sural nerve cross-sectional area determined by ultrasound in oxaliplatin-induced peripheral neuropathy patients will be transformed to compare to historical data previously collected from healthy adults and oxaliplatin-induced peripheral neuropathy patients using analysis of variance (ANOVA).
Amplitude of Nerve Response of Tibial Nerve | Up to 30 days
  Amplitude will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
Amplitude of Nerve Response of Sural Nerve | Up to 30 days
  Amplitude will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
Distal Latency of Nerve Response of Tibial Nerve | Up to 30 days
  Distal latency will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
Distal Latency of Nerve Response of Sural Nerve | Up to 30 days
  Distal latency will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
Conduction Velocity of Nerve Response of Tibial Nerve | Up to 30 days
  Conduction velocity will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
Conduction Velocity of Nerve Response of Sural Nerve | Up to 30 days
  Conduction velocity will be obtained from a nerve conduction study. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and nerve conduction studies.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (EORTC QLQ-CIPN20) Questionnaire | Up to 30 days
  A 20-item self-reported neuropathy score questionnaire for participants to report neuropathy symptoms or problems. Scoring ranges from 1-4, 1 being not at all, 4 being very much.
Reduction of Intraepidermal Nerve Fiber Density | Up to 30 days
  Biopsies will be taken from the distal leg or proximal thigh to evaluate peripheral neuropathy. Spearman's rank correlation coefficient will be used to examine the associations between nerve cross-sectional area and intraepidermal nerve fiber density.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03958747/ICF_000.pdf